CLINICAL TRIAL: NCT03091322
Title: BIO|MASTER.Edora Family Study
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: BA106
Record Dates: First submitted 2017-01-27; First posted 2017-03-27 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-01

CONDITIONS: Pacemaker Therapy; Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SR-T group: single chamber pacemaker
  Interventions: Device: Pacemaker of the Edora Family (Edora/ Evity/ Enitra/ Enticos) 8
- DR-T group: dual chamber pacemaker
  Interventions: Device: Pacemaker of the Edora Family (Edora/ Evity/ Enitra/ Enticos) 8
- HF-T group: triple chamber pacemaker (IS-1 connector)
  Interventions: Device: Pacemaker of the Edora Family (Edora/ Evity/ Enitra/ Enticos) 8
- HF-T QP group: triple chamber pacemaker (with IS4 connector) and a lead of the Sentus QP lead family
  Interventions: Device: Pacemaker of the Edora Family (Edora/ Evity/ Enitra/ Enticos) 8

INTERVENTIONS:
Device: Pacemaker of the Edora Family (Edora/ Evity/ Enitra/ Enticos) 8 — Assessment of the AV Opt and LV VectorOpt features

SUMMARY:
This study is designed as post market clinical follow-up study with CE-marked products to evaluate the AV Opt and LV VectorOpt features in the respective Edora family pacemakers under clinical conditions. Furthermore, adverse events will be evaluated to identify residual risks associated with the use of the BIOTRONIK Edora family pacemakers. The study is further designed to address potential regulatory needs of clinical data for countries and regions not covered by the CE approval.

DETAILED DESCRIPTION:
Study Design

* Open-label, prospective, non-randomized, multicenter, international
* about 13 study sites

Study Endpoints

The following endpoints are defined and will be assessed with descriptive analysis:

1. AV Opt feature:

   The feature's AV delay recommendation was
   1. used as basis for the device programming or is at least considered to be clinically acceptable or
   2. other AV delay values were chosen by the investigator and the recommendation was rated as not clinically acceptable.
2. LV VectorOpt usability using an overall score (categories: excellent, good, average, fair, poor).
3. (S)ADEs and calculation of the SADE free rate until the 6-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for pacemaker therapy or cardiac resynchronization therapy
* Patient is able to understand the nature of the study;
* Patient provides written informed consent;
* Patient is able and willing to complete the planned follow-up visits at the investigational site;
* Patient accepts Home Monitoring® concept;
* Age ≥ 18 years.

Exclusion Criteria:

* Any contraindication for pacemaker or cardiac resynchronization therapy (whichever applies);
* Patient has received or is planned to receive an epicardial LV lead implant;
* Pregnant or breast-feeding;
* Life expectancy of less than 6 months;
* Participation in an interventional clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for cardiac pacemaker or cardiac resynchronization therapy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
AV delay recommendation by the AV Opt Feature was either used for the device programming or was rated as clinically acceptable. | until the 1-month follow-up
  The AV Opt Feature will be assessed only for patients with triple-chamber devices and patients with dual-chamber devices (if clinically indicated) with sinus rhythm of sufficient intrinsic rate. According to the clinical investigation plan this endpoint will be assessed with descriptive analysis methods.
Overall score for the usability of the LV VectorOpt feature | until the 1-month follow-up
  The LV VectorOpt feature has to be assessed for patients with an HF-T device (triple-chamber) and a QP lead (quadripolar, HF-T QP group) only. According to the clinical investigation plan this endpoint will be assessed with descriptive analysis methods.
(S)ADEs and calculation of the SADE free rate | until the 6-month follow-up
  Descriptive analysis of all (S)ADEs and calculation of the SADE free rate

CONTACTS AND LOCATIONS:
Locations (11):
- Kepler Universitätsklinikum, Linz, Austria
- Germany (8):
  - Maria Heimsuchung - Caritas-Klinik Pankow, Berlin
  - Herzzentrum Bernau, Bernau
  - Städtisches Klinikum Brandenburg GmbH, Brandenburg
  - Klinikum St. Georg gGmbH, Leipzig
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Niels-Stensen-Kliniken, Marienhospital Osnabrück, Osnabrück
  - Universitätsklinikum Würzburg, Würzburg
  - Heinrich-Braun-Klinikum gemeinnützige GmbH, Zwickau
- Clínica Universitaria de Navarra (CUN), Pamplona, Spain
- Luzerner Kantonsspital (LUKS), Lucerne, Switzerland